CLINICAL TRIAL: NCT02934802
Title: Non-Interventional Consecutive and Prospective Study of e.Motion® PS Pro Prosthesis in the Total Knee Artroplasty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: BBraun Medical SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1420
Record Dates: First submitted 2016-10-14; First posted 2016-10-17 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Knee Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Total Knee prothesis e motion PS Pro

SUMMARY:
This post-market clinical follow-up study intends to investigate the survival rate at 5 years of the e.motion® PS Pro System.

ELIGIBILITY:
Inclusion Criteria:

* Patient having signed informed consent
* Patients over 18 for which a Total Knee Prosthesis with e.motion® PS Pro was decided
* Patients willing to participate in a 5 years follow-up

Exclusion Criteria:

* Active or suspected infection
* Tumor on the concerned knee
* Patient vulnerable and under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients for which a Total Knee Prosthesis with e.motion® PS Pro was decided by the surgeon
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2016-05-26 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Survival rate at 5 years of the e motion PS Pro | the survival rate will be evaluated 6-12 weeks; 1; 2; 3; 4 and 5 years after the knee arthroplasty
  The endpoint is the revision of at least one of the prosthesis components. If a patient withdraws from the study for any reason, counts as the end date for the survival of the implant of the last day on which the implants were well known even in place.

CONTACTS AND LOCATIONS:
Overall Officials: François Boillot, Principal Investigator — Groupe hospitalier Paris-St Joseph
Locations (1):
- Groupe hospitalier Paris-St Joseph, Paris, France

IPD SHARING:
Plan to Share IPD: No